CLINICAL TRIAL: NCT05561491
Title: An Open-Label, Two-Part, Dose-Exploration and Multiple Expansion, Phase 2 Study of ONCOS-102 in Combination With Novel Immune-Targeted Anti-Cancer Agents in Patients With Unresectable or Metastatic Cutaneous Melanoma Resistant to Anti-PD-(L)1 Treatment
Brief Title: A Study of ONCOS-102 in Combination With Other Novel Immune-therapies in Advanced Treatment-resistant Melanoma Patients
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Strategic reasons
Sponsor: Targovax Oy (Industry)
Collaborators: Agenus Inc. (Industry)
Responsible Party: Sponsor
Organization: Targovax ASA (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOPHOS-213
Record Dates: First submitted 2022-09-27; First posted 2022-09-30 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-05

CONDITIONS: Melanoma
Keywords: ONCOS-102; balstilimab; checkpoint inhibitor; oncolytic virus; PD-1; PD-L1; refractory; metastatic
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis | interventions — balstilimab

STUDY DESIGN:
Intervention Model Description: 2 part dose escalation and multiple expansion phase 2 trial.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ONCOS-102 (Experimental): ONCOS-102 will be administered by intratumoral (IT) injection at 1.0×10^12 VP/dose with the potential to de-escalate dosing to 3.0×10^11 VP/dose.
  Interventions: Biological: ONCOS-102
- ONCOS-102 and balstilimab (Experimental): ONCOS-102 will be administered by IT injection at 3.0×10^11 VP/dose with planned dose escalation to 1.0×10^12 VP/dose. Balsitilmab will be administered at a fixed dose of 300 mg by intravenous (IV) injection.
  Interventions: Biological: ONCOS-102; Biological: Balstilimab

INTERVENTIONS:
Biological: ONCOS-102 — Oncolytic virus
Biological: Balstilimab — Anti PD-1
  Arms: ONCOS-102 and balstilimab

SUMMARY:
A Phase 2 study investigating the efficacy and safety of ONCOS-102 alone or in combination with balstilimab (a programmed death receptor-1 [PD-1] inhibitor).

DETAILED DESCRIPTION:
This study will test ONCOS-102 in combination with novel immune-targeted anti-cancer agents in patients with unresectable or metastatic cutaneous melanoma resistant to anti-PD (L)1 treatment. The purpose of this study is to further evaluate safety and tolerability, as well as anti-tumour activity of ONCOS-102 (both as monotherapy and in combination with anti-PD-1 balstilimab) in the target population.

Following a safety run-in period, up to approximately 63 participants with cutaneous melanoma who previously progressed on anti-PD-1/L1-based therapy will be allocated 1:1 to receive either ONCOS-102 alone or ONCOS-102 plus balstilimab.

Part 1 - Dose Exploration Run-in: Part 1 of the study will evaluate and further optimise the dose of ONCOS-102; a recommended phase 2 dose (RP2D) for ONCOS-102 will be identified.

Part 2 - Multiple Expansion: In the expansion phase, ONCOS-102 alone or in combination with balstilimab will be further evaluated in Cohorts 1 and 2 using the RP2D identified in Part 1.

The study is structured to allow for additional combination cohorts to be added to the study following a protocol amendment.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent for the study.
2. Be ≥ 18 years of age on the day of signing the informed consent form (ICF).
3. Eastern Co-operative Oncology Group (ECOG) performance status 0 or 1.
4. Histologically confirmed diagnosis of metastatic or unresectable malignant melanoma at screening with measurable disease (by RECIST v1.1) that is accessible for IT injection into cutaneous or subcutaneous lesions.
5. Resistant to PD-(L)1 blockade (primary or secondary resistance in the advanced setting or relapse after adjuvant therapy) either as monotherapy or in combination with other therapies, as defined by the following criteria:

   * Received at least 1 prior anti-PD-[L]1 immunotherapy regimen for a minimum of 6 weeks.
   * Prior progression must be either on treatment with anti-PD-(L)1 or ≤ 12 weeks from last dose in metastatic setting or relapse ≤ 24 weeks from completion of therapy in adjuvant setting.
   * Has demonstrated disease progression (PD) after anti-PD-(L)1 as defined by RECIST v1.1. The initial evidence of PD is to be confirmed by a second assessment (i.e., a confirmatory scan no less than 4 weeks from the date of the first documented PD), in the absence of clear clinical progression.
6. Has recovered from all adverse events (AEs) due to previous therapies to ≤ Grade 1 or baseline. Patients with ≤ Grade 2 endocrinopathies stable on mediation, stable neuropathy, and alopecia are eligible.

Exclusion Criteria:

1. Uveal or mucosal melanoma.
2. Any history of National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Grade ≥ 3 immune-mediated toxicity (excluding endocrinopathies and non-necrotising/bullous rash) from prior checkpoint inhibition.

   • If prior severe toxicity occurred during combination treatment with anti-PD-(L)1 + anti-cytotoxic lymphocyte associated antigen 4 (CTLA-4) but subsequent treatment with anti-PD-(L)1 as monotherapy was tolerated, the patient may be eligible for inclusion after discussion with the medical monitor.
3. Has known (current or previously treated) central nervous system metastases and/or carcinomatous meningitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events [safety and tolerability] of ONCOS-102 monotherapy and ONCOS-102 plus balstilimab. | 90 days after last treatment
  To determine the incidence of treatment emergent adverse events including treatment emergent serious adverse events assessed by CTCAE v5.0, treatment interruptions and discontinuations.
To evaluate the objective response rate (ORR) in individual cohorts using RECIST v1.1 | Up to 27 months after the last patient first dose
  The proportion of patients achieving confirmed complete (CR) or partial response (PR) per RECIST v1.1 criteria

SECONDARY OUTCOMES:
To evaluate the duration of response (DoR) in individual cohorts | Up to 27 months after the last patient first dose
  Time from observed objective response to first occurrence of disease progression or death based on Investigator assessment according to RECIST v1.1
To evaluate progression-free survival (PFS) in the individual cohorts using the Kaplan-Meier method | Up to 27 months after last patient recruited per cohort
  Time from treatment initiation to first occurrence of disease progression or death based on Investigator assessment according to RECIST v1.1
To evaluate overall survival (OS) in individual cohorts using the Kaplan-Meier method | Up to 27 months after last patient recruited per cohort
  Time from treatment initiation to death that occurred up to 24 months after the last patient recruited per cohort
To evaluate PFS rate estimates at 3, 6 and 12 months in individual cohorts | 3, 6 and 12 months after last patient recruited per cohort
  Proportion of patients with a partial or complete response to treatment observed at Month 3 (Month 6 and Month 12) based on RECIST v1.1
To evaluate systemic exposure of ONCOS-102 | Up to 24 months after last patient in the PK sampling group
  Concentration of virus particles in blood and non-compartmental PK parameters as data allow.
To estimate baseline presence and incidence of ONCOS-102 anti-drug antibodies (ADA) and neutralising antibodies (NAb) during study | Up to 24 months after last patient in the pharmacokinetic sampling group
  ADA (screening, confirmatory results: positive or negative; titres), NAb (titres)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas B Johnson, MD, MSCI, Principal Investigator — Vanderbilt Institute for Infection, Immunology and Inflammation